CLINICAL TRIAL: NCT05828342
Title: Use of the Loss-of-resistance Syringe Technique in Determining Endotracheal Cuff Measurements in Pediatric Patients
Brief Title: Loss-of-resistance Syringe Technique in Determining Endotracheal Cuff Pressure
Status: Completed | Type: Observational
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Yusuf Yılmaz, Specialist Physician, Ankara City Hospital Bilkent
Other Study IDs: E2-22-2060
Record Dates: First submitted 2023-04-12; First posted 2023-04-25 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Endotracheal Tube Cuff Pressure; Loss of Resistance Syringe; Airway Edema; Pediatric Population
Keywords: Airway; Cuff Pressure; Endotracheal Tube

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric Patients: Patients under the age of 18 who were operated under general anesthesia and intubated with a cuffed endotracheal tube between 15 July 2022 and 15 October 2022 in the pediatric operating room.
  Interventions: Procedure: Endotracheal tube cuff inflation with the loss of resistance syringe method

INTERVENTIONS:
Procedure: Endotracheal tube cuff inflation with the loss of resistance syringe method — The cuffs of the endotracheal tubes will be inflated with the epidural loss of resistance syringe, the syringe piston will be released, the syringe piston will be pushed back with oscillation, and then the cuff pressures will be measured and recorded with a cuff manometer (VBM Cuff Pressure Gauge) and an electronic injector that measures cuff pressure (AG Cufill). A three-way vein valve will be used when making this measurement. During the measurement, an epidural resistance loss injector will be attached to one valve, a cuff manometer attached to another valve, and an electronic injector (AG Cufill) measuring cuff pressure to the third track. With this technique, the possibility of leakage due to insertion and removal during measurements will be eliminated.

SUMMARY:
The goal of this observational study is to learn about whether the loss-of-resistance syringe technique is beneficial when adjusting endotracheal cuff pressure in pediatric patients.

The main questions it aims to answer are:

* Is the loss of resistance syringe technique useful when adjusting endotracheal cuff pressure in pediatric patients?
* Is there a difference between the measurements of two different cuff manometers used in the clinic, if so, what is the safety margin between the two manometers?

The participants who will be operated under general anesthesia will be anesthetized with the standard anesthesia method, the cuffs of the endotracheal tubes will be inflated with an epidural loss of resistance syringe, the syringe piston will be released, and then the syringe piston will be pushed back with oscillation. Then, cuff pressures will be measured and recorded with a cuff manometer (VBM Cuff Pressure Gauge) and an electronic injector measuring cuff pressure (AG Cufill).

DETAILED DESCRIPTION:
Various complications related to endotracheal tube may develop after general anesthesia. Inflated cuffs at inappropriately high pressure reduce tracheal mucosal blood flow, causing ischemia and tracheal stenosis in the future. Cuffs that are inflated at lower pressures than necessary can cause inadequate ventilation and aspiration of stomach contents. Adequate endotracheal cuff pressure should be between 20-30 cmH2O. Cuff pressure should be kept around 25 cmH2O in critically ill intubated and mechanically ventilated patients. In critically ill patients, such as intensive care patients, contaminated secretions can leak from the tracheal cuff and cause ventilator-associated pneumonia. High cuff pressure increases the risk of tracheomalacia and tracheal dilatation in patients who are intubated for a long time.

Inflating the endotracheal cuff at the correct pressure is the main precaution in preventing complications such as tracheal stenosis. Cuff manometers are manual or automatic devices that measure pressure in endotracheal tube (ETT) or laryngeal mask airway (LMA) cuffs, and some may operate to maintain pressure at a certain level for extended periods of time. However, it is not always possible to understand that the endotracheal cuff is inflated at the correct pressure due to operating room insufficiencies. Not every operating room has a cuff manometer, and various manual techniques are used by anesthesiologists to inflate the endotracheal cuff without a cuff manometer. One of these techniques is the palpation technique applied by experienced anesthesiologists. However, this technique is known to have a high rate of errors. It has been shown that professional experience does not contribute to achieving the correct cuff pressure without pressure monitoring. Another technique is the "loss of resistance syringe technique". It aims to equalize the endotracheal cuff pressure to the tracheal lateral wall pressure by releasing the syringe piston after inflating the endotracheal cuff with a loss of resistance syringe, allowing the air pressure inside the cuff to push the syringe piston passively. This technique has been used previously in adult patients and has been proposed as an economical and easily accessible method for inflating the endotracheal cuff. There is no study in the literature on the use of this technique in pediatric patients.

In this study, investigators aimed to find out whether the resistance loss syringe technique is useful when adjusting the endotracheal cuff pressure in pediatric patients. Secondary aim of the study is to evaluate the measurements of two different manometers and to determine the margin of safety between the two manometers.

Benefit from research; the aim is to facilitate the inflation of the endotracheal cuffs of pediatric patients intubated under general anesthesia at the correct pressure and to prevent possible complications. The study does not have any risks other than possible general anesthesia risks.

This study is a clinical observational prospective study. Participants were patients between the ages of 0-18 who were anesthetized with standard general anesthesia method in the pediatric operating room and intubated with a cuffed endotracheal tube. Then, the cuff of the endotracheal tubes will be inflated with the epidural loss of resistance syringe, after that the syringe piston will be released, the syringe piston will be pushed back by the cuff pressure, and then the cuff pressures will be measured and recorded with the cuff manometer (VBM Cuff Pressure Gauge) and the cuff pressure measuring electronic injector (AG Cufill). A three-way vein valve will be used when making this measurement. During the measurement, an epidural loss of resistance syringe will be attached to one valve, a cuff manometer attached to another valve, and an electronic injector (AG Cufill) measuring cuff pressure to the third track. With this technique, the possibility of leakage due to insertion and removal during measurements will be eliminated. The tube number of the patients will be determined according to the age-based formula and according to the anesthetist's prediction during intubation. Then it will be checked whether there is an air leak in the mechanical ventilator. The endotracheal tube cuff of patients with airway leakage will be inflated under the guidance of the cuff manometer so that there is no leakage.

ELIGIBILITY:
Inclusion Criteria:

-Patients under the age of 18 who will be intubated and operated under general anesthesia in the pediatric operating room, whose informed consent form has been approved by their parents, between July 15, 2022 and October 15, 2022

Exclusion Criteria:

- Patients who are considered for difficult intubation, trachamalacia, laryngomalacia, tracheal surgery, or whose parental consent form has not been approved will be excluded from the study.

Max Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Pediatric Population
Sampling Method: Probability Sample
Enrollment: 198 (Actual)
Dates: Start 2022-07-15 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-10-15 (Actual)

PRIMARY OUTCOMES:
Pressure of the cuff inflated with the loss-of-resistance syringe technique | 1 minute
  The primary outcome is to find out whether the loss-of-resistance syringe technique is beneficial when adjusting endotracheal cuff pressure in pediatric patients. With this technique, it will be checked whether the cuff pressures inflated are between 20-30 cm H2O. Endotracheal cuff pressure will be recorded with manometer.
Percentage of airway leak | 1 minute
  After the patients' endotracheal cuffs are inflated with a loss of resistance syringe, the mechanical ventilator will be checked for airway leakage. If there is a leak, the percentage of the leak will be recorded.

SECONDARY OUTCOMES:
Pressure difference between different types of manometers | 1 minute
  The secondary aim of the study is to evaluate the measurements of two different manometers used in the clinic and to determine the margin of safety between the two manometers. Endotracheal cuff pressure will be recorded with two different manometers.

CONTACTS AND LOCATIONS:
Overall Officials: Sengul Ozmert, Study Director — Ankara CH Bilkent; Ayça T Dumanlı Ozcan, Study Director — Ankara CH Bilkent
Locations (1):
- Ankara City Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Nseir S, Brisson H, Marquette CH, Chaud P, Di Pompeo C, Diarra M, Durocher A. Variations in endotracheal cuff pressure in intubated critically ill patients: prevalence and risk factors. Eur J Anaesthesiol. 2009 Mar;26(3):229-34. doi: 10.1097/eja.0b013e3283222b6e. PMID 19244697
- [Background] Weiss M, Doell C, Koepfer N, Madjdpour C, Woitzek K, Bernet V. Rapid pressure compensation by automated cuff pressure controllers worsens sealing in tracheal tubes. Br J Anaesth. 2009 Feb;102(2):273-8. doi: 10.1093/bja/aen355. Epub 2008 Dec 25. PMID 19112060
- [Background] Dubey M, Kumar Mittal A, Choudhary M. Loss of Resistance Syringe: A Substitute for Cuff Pressure Manometer. Anesth Analg. 2017 Aug;125(2):701-703. doi: 10.1213/ANE.0000000000002235. No abstract available. PMID 28737520